CLINICAL TRIAL: NCT01809132
Title: Double-blind Randomized Controlled Trial of Anakinra, Pentoxifylline, and Zinc Compared to Methylprednisolone in Severe Acute Alcoholic Hepatitis
Brief Title: Efficacy Study of Anakinra, Pentoxifylline, and Zinc Compared to Methylprednisolone in Severe Acute Alcoholic Hepatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mack Mitchell (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); The Cleveland Clinic (Other); University of Massachusetts, Worcester (Other); University of Louisville (Other)
Responsible Party: Sponsor-Investigator, Mack Mitchell, Professor of Medicine, Division of Digestive and Liver Diseases, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01AA021893-01 (NIH); U01AA021893-01 (NIH)
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Acute Alcoholic Hepatitis
Keywords: Hepatitis, alcoholic; pentoxifylline; zinc; anakinra; glucocorticoids; MELD score; Intestinal mucosa
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Interleukin 1 Receptor Antagonist Protein; Pentoxifylline; Drugs, Generic; Zinc Sulfate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anakinra & Pentoxifylline & Zinc Sulfate (Experimental): anakinra 100mg subcutaneous injection daily for 14 days pentoxifylline 400 mg orally three times daily for 28 day zinc sulfate 220 mg orally for 180 days
  Interventions: Drug: Anakinra; Drug: Pentoxifylline; Drug: Zinc Sulfate
- Methylprednisolone (Active Comparator): methylprednisolone 32 mg orally daily for 28 days
  Interventions: Drug: Methylprednisolone
- Observational (No Intervention): Individuals who choose not to participate in the interventional arm of the trial will be receive standard care and be observed for 6 months. They will be enrolled to have baseline and interval health information and laboratory results collected.

INTERVENTIONS:
Drug: Anakinra — Anakinra, interleukin-1 receptor antagonist; 100 mg/0.67 mL solution for subcutaneous injection.
  Other Names: Kineret
  Arms: Anakinra & Pentoxifylline & Zinc Sulfate
Drug: Pentoxifylline — Pentoxifylline, generic
  Other Names: Pentoxifylline, generic
  Arms: Anakinra & Pentoxifylline & Zinc Sulfate
Drug: Zinc Sulfate — Zinc Sulfate, nutritional supplement
  Other Names: Zinc Sulfate, generic
  Arms: Anakinra & Pentoxifylline & Zinc Sulfate
Drug: Methylprednisolone — Methylprednisolone, corticosteroid
  Other Names: Methylprednisolone, generic
  Arms: Methylprednisolone

SUMMARY:
This study will compare two different treatments of acute alcoholic hepatitis. The current standard of care is treatment with corticosteroids (methylprednisolone). This will be compared to treatment with anakinra, pentoxifylline, plus zinc sulfate. The participants will be treated and followed for 6 months and the two treatment groups will be compared for differences in death rates and laboratory tests that measure liver and gut function.

DETAILED DESCRIPTION:
This study will test the hypothesis that the syndrome of acute alcoholic hepatitis results from severe inflammation and dysregulated cytokines. Steroid monotherapy is not effective in all patients and this study will utilize compounds that have the potential to improve gut barrier function, to reduce the associated inflammation, and to prevent the development of hepatorenal syndrome and other organ failure.

Patients will be randomized to receive 28 days of methylprednisolone 32 mg daily OR therapy that includes a combination of anakinra (interleukin-1 receptor antagonist) 100mg by subcutaneous injection daily for 14 days plus pentoxifylline 400 mg orally three times daily for one month plus zinc supplements (220 mg of zinc sulfate) given orally for 6 months. This combination strategy will address the acute inflammatory component of the disease (anakinra) and protect against development of hepatorenal syndrome (pentoxifylline), one of the most frequent causes of death in severe acute alcoholic hepatitis, and improve gut mucosal integrity (zinc supplements). The primary outcome will be 6 month mortality rate. Secondary outcomes will be measured at 30, 90 and 180 days.

Individuals who are not participating in the interventional arm of the trial will be receive standard care and be observed for 6 months. They will be enrolled to have baseline and interval health information and laboratory results collected.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent by subject or appropriate family member
2. Age between 21-70 years
3. Recent alcohol consumption > 50 g/d for > 6 months, continuing within two months before enrollment
4. d. At least 2 of the following symptoms of acute alcoholic hepatitis: Anorexia, nausea, RUQ pain
5. Liver biopsy showing alcoholic hepatitis (steatohepatitis) OR ultrasound of liver showing increased echogenicity OR CT scan showing decreased attenuation of liver compared to spleen OR MRI showing fatty liver (decreased signaling intensity on T1 weighted images) If liver biopsy confirms diagnosis of alcoholic hepatitis then requirement for AST elevation > 50 is waived. The liver biopsy must be done within 60 days of study enrollment.
6. AST levels:

   * AST> Or equal to 50 IU/mL but less than 500 IU/mL
   * AST> ALT, ratio AST/ALT> 1.5; ALT < 200 IU/mL
   * or biopsy proven alcoholic hepatitis.
7. Model for End-Stage Liver Disease (MELD) ≥ 20 and Maddrey DF ≥ 32.
8. Willingness to utilize two reliable forms of contraception (both males and females of childbearing potential) from screening through the first 6 weeks of the study.

Exclusion Criteria:

1. Hypotension with BP < 80/50 after volume repletion
2. Pregnancy; incarceration; inability to provide consent or lack of appropriate family member
3. Signs of uncontrolled systemic infection: Fever > 38°C and positive blood or ascites cultures and on appropriate antibiotic therapy for ≥ 3 days within 3 days of inclusion
4. Acute gastrointestinal bleeding requiring >2 units blood transfusion within the previous 4 days
5. Undue risk from immunosuppression: Positive HBsAg; a positive skin PPD skin test, a positive quantiferon, or history of treatment for tuberculosis; history of any malignancy except skin cancer but including hepatocellular carcinoma within the last five years; HIV infection
6. Recent previous treatment with corticosteroids or other immunosuppressive medications including specific anti-TNF therapy (not including pentoxifylline), calcineurin inhibitors within the previous 3 months. Treatment with corticosteroids for ≤3 days prior to baseline is acceptable.
7. Evidence of acute pancreatitis: CT evidence or amylase or lipase > 5 X upper limit of normal (ULN).
8. Serious cardiac, respiratory or neurologic disease or evidence of other liver diseases such as autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson disease, hemochromatosis, secondary iron overload due to chronic hemolysis, alpha-1-antitrypsin deficiency
9. Acute or chronic kidney injury with serum creatinine > 3.0 mg/dl.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mack C Mitchell, MD, Principal Investigator — University of Texas Southwestern Medical Center; Arthur J McCullough, MD, Principal Investigator — The Cleveland Clinic; Craig J McClain, MD, Principal Investigator — University of Louisville; Gyongi Szabo, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (4):
- United States (4):
  - University of Louisville, Louisville, Kentucky
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Hassanein T, McClain CJ, Vatsalya V, Stein LL, Flamm SL, Martin P, Cave MC, Mitchell M Jr, Barton B, Nagy L, Szabo G, McCullough A, Dasarathy S, Shah J, Blevins C, Scott D, Krebs W, Brown JE, Lin W. Safety, Pharmacokinetics, and Efficacy Signals of Larsucosterol (DUR-928) in Alcohol-Associated Hepatitis. Am J Gastroenterol. 2024 Jan 1;119(1):107-115. doi: 10.14309/ajg.0000000000002275. Epub 2023 Apr 3. PMID 37011138
- [Derived] Szabo G, Mitchell M, McClain CJ, Dasarathy S, Barton B, McCullough AJ, Nagy LE, Kroll-Desrosiers A, Tornai D, Min HA, Radaeva S, Holbein MEB, Casey L, Cuthbert J. IL-1 receptor antagonist plus pentoxifylline and zinc for severe alcohol-associated hepatitis. Hepatology. 2022 Oct;76(4):1058-1068. doi: 10.1002/hep.32478. Epub 2022 Jun 2. PMID 35340032
- [Derived] Helsley RN, Miyata T, Kadam A, Varadharajan V, Sangwan N, Huang EC, Banerjee R, Brown AL, Fung KK, Massey WJ, Neumann C, Orabi D, Osborn LJ, Schugar RC, McMullen MR, Bellar A, Poulsen KL, Kim A, Pathak V, Mrdjen M, Anderson JT, Willard B, McClain CJ, Mitchell M, McCullough AJ, Radaeva S, Barton B, Szabo G, Dasarathy S, Garcia-Garcia JC, Rotroff DM, Allende DS, Wang Z, Hazen SL, Nagy LE, Brown JM. Gut microbial trimethylamine is elevated in alcohol-associated hepatitis and contributes to ethanol-induced liver injury in mice. Elife. 2022 Jan 27;11:e76554. doi: 10.7554/eLife.76554. PMID 35084335
- [Derived] Vatsalya V, Cave MC, Kong M, Gobejishvili L, Falkner KC, Craycroft J, Mitchell M, Szabo G, McCullough A, Dasarathy S, Radaeva S, Barton B, McClain CJ. Keratin 18 Is a Diagnostic and Prognostic Factor for Acute Alcoholic Hepatitis. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2046-2054. doi: 10.1016/j.cgh.2019.11.050. Epub 2019 Dec 4. PMID 31811953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational
Started | 53 | 50 | 1 (Subject was consented but withdrew prior to randomization and initiation of treatment.)
Completed | 53 | 50 | 0
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational | Total
Number analyzed (Participants) | 53 | 50 | 1 | 104
Age, Categorical [Count of Participants; unit: Participants] — Population: The observational subject was lost to follow up.
  Participants
    number analyzed (Participants) | 53 | 50 | 0 | 103
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 53 | 50 | 0 | 103
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 1 | 41
  Male | 35 | 28 | 0 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 0 | 19
  Not Hispanic or Latino | 38 | 38 | 1 | 77
  Unknown or Not Reported | 5 | 3 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 0 | 8
  White | 47 | 47 | 1 | 95
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 180 Days Mortality
Description: Death at 180 days
Time Frame: Time to event up to 6 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational
Number analyzed (Participants) | 53 | 50 | 0
Participants | 17 | 22 | 0
Statistical Analysis 1: Comparison: Anakinra & Pentoxifylline & Zinc Sulfate vs Methylprednisolone; Test type: Superiority; p = .30, Log Rank

2. Secondary Outcome: MELD Score at 28 Days
Description: Model of End Stage Liver Disease Score calculated from serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR). MELD score ranges from 6-40. A higher score indicates a lesser outcome.
  The Model for End Stage Liver Disease scoring system is based on the INR, total serum bilirubin and serum creatinine. The measure reflects 90 day prognosis of alcohol associated liver disease from the time of measurement and therefore can only be assessed on subjects who are alive at the specified time point since lab values from that time point are required for the measure.
Time Frame: 28 days
Population: This outcome could not be calculated for the observational subject who was lost to follow up.
  Analysis were limited to the subjects that were alive for this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational
Number analyzed (Participants) | 30 | 29 | 0
score on a scale | 22.57 (6.31) | 20.95 (6.44) |
Statistical Analysis 1: Comparison: Anakinra & Pentoxifylline & Zinc Sulfate vs Methylprednisolone; the observational subject was lost to follow-up; Test type: Superiority; p = .42, t-test, 2 sided

3. Secondary Outcome: MELD Score at 90 Days
Description: as for outcome 2
Time Frame: 90 Days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational
Number analyzed (Participants) | 22 | 17 | 0
score on a scale | 15.50 (6.11) | 16.38 (9.58) |
Statistical Analysis 1: Comparison: Anakinra & Pentoxifylline & Zinc Sulfate vs Methylprednisolone; Test type: Superiority; p = .75, t-test, 2 sided

4. Secondary Outcome: MELD Score at 180 Days
Description: as for outcome 2
Time Frame: 180 Days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational
Number analyzed (Participants) | 19 | 15 | 0
score on a scale | 15.81 (10.10) | 11.85 (4.47) |
Statistical Analysis 1: Comparison: Anakinra & Pentoxifylline & Zinc Sulfate vs Methylprednisolone; Test type: Superiority; p = .17, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definitions of adverse events are the same as those used in clinicaltrials.gov Adverse events were not collected for the observational arm.
Groups:
- Observational: Individuals who choose not to participate in the interventional arm of the trial will receive standard care and be observed for 6 months. They will be enrolled to have baseline and interval health information and laboratory results collected.
Arm/Group | Anakinra & Pentoxifylline & Zinc Sulfate | Methylprednisolone | Observational
All-Cause Mortality (participants affected / at risk) | 17/53 | 22/50 | 0/0
Serious Adverse Events (participants affected / at risk) | 33/53 | 30/50 | 0/0
Other Adverse Events (participants affected / at risk) | 20/53 | 4/50 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra & Pentoxifylline & Zinc Sulfate (N=53) | Methylprednisolone (N=50) | Observational (N=0)
Acute Kidney Injury (Renal and urinary disorders) | 10 (10) | 13 (13) | 0 (0)
Upper GI hemorrhage (Vascular disorders) | 4 (4) | 4 (4) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Nocardia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Histoplasmosis infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Baceteremia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Multiple Organ Dysfunction Syndrome (MODS) (General disorders) | 2 (2) | 3 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Esophageal varices hemorrhage (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Ascites (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra & Pentoxifylline & Zinc Sulfate (N=53) | Methylprednisolone (N=50) | Observational (N=0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0)
Hematemesis (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Ascites (Hepatobiliary disorders) | 3 (3) | 3 (3) | 0 (0)
C. difficile infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT01809132/Prot_SAP_000.pdf